CLINICAL TRIAL: NCT06301139
Title: Clinical Trial to Assess Improvement of Digestive Symptoms With Goat's Milk Infant Formula.
Brief Title: Goat Milk Infant Formula Comfort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ausnutria Hyproca B.V. (Industry)
Collaborators: HM hospitales (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P17-004
Record Dates: First submitted 2024-02-28; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Gastrointestinal Diseases; Cow's Milk Intolerance
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: randomized controlled pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goat milk-based formula (Experimental): goat milk-based infant formula (GMF)
  Interventions: Dietary Supplement: Goat milk-based infant formula
- Cow's milk-based formula (Placebo Comparator): cow's milk-based infant formula supplemented with probiotics (CMFp)
  Interventions: Dietary Supplement: Cow's milk-based infant formula with probiotic drops

INTERVENTIONS:
Dietary Supplement: Goat milk-based infant formula — Infant formula based on goat milk for 4 weeks at volume depending on the infant
  Arms: Goat milk-based formula
Dietary Supplement: Cow's milk-based infant formula with probiotic drops — Infant formula based on cow's milk with probiotic Lactobacillus reuteri drops for 4 weeks at volume depending on the infant
  Arms: Cow's milk-based formula

SUMMARY:
In this study, the investigators aim to assess that infants with mild symptoms have significantly less (severe) symptoms after 14 days goat milk-based formula use compared to infants using cow's milk-based formula supplemented with probiotic drops.

DETAILED DESCRIPTION:
Anecdotal evidence shows that the use of goat milk-based infant formula decreases discomfort of infants with cow's milk related symptoms. In this randomized controlled pilot study, the effect on comfort during usage of goat-milk based infant formula is studied. Twenty formula fed infants (aged between 6 weeks and 3 months) who experience mild discomfort will receive goat milk-based infant formula (GMF) or cow's mik based infant formula supplemented with probiotics lactobacillus reuteri drops (CMFp). The infants will be assessed by a local paediatricians using the Cow's Milk-related Symptom Score (CoMiSS). This is a fast, non-invasive and easy-to-use and validated questionnaire to assess infant's reaction to proteins found in cow's milk. The higher the score, the more sensitive the child is to cow's milk proteins, the maximum score is 33 points. Infants with a CoMiSS Score between 6 and 12 will be enrolled in this study. It is expected that infants will have a better response to GMF, which will result in a decrease of the CoMiSS Score after a 2 weeks intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy full-term infant with birth weight ≥2,500 to ≤4,500 g
* Infant aged between 4 weeks and 3 months at enrolment
* CoMiSS value at baseline between 6 and 12
* Infant is exclusively bottle fed with cow's milk based infant formula at baseline

Exclusion Criteria:

* Breastfed infants
* Congenital illness or malformation that may affect infant feeding or normal growth
* Gastrointestinal disorders
* Confirmed cow or goat milk protein allergy or lactose intolerance
* Supplemental feeding
* Readmission to hospital for longer than 3 days for another reason than hyperbilirubinemia prior to enrolment
* Infant participating in another clinical study

Ages: 6 Weeks to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Cow's Milk-related Symptoms | 0-2 weeks
  Difference in Cow's Milk related Symptom Score (CoMiSS: score ranges from 0 to 33 with higher scores indicating more symptoms) at baseline and after 14 days of intervention.

SECONDARY OUTCOMES:
Cow's Milk-related Symptoms | 0-4 weeks
  Difference in Cow's Milk-related Symptoms Score (CoMiSS: score ranges from 0 to 33 with higher scores indicating more symptoms) at baseline and after 28 days of intervention.
Parental stress | 0-4 weeks
  Difference in parental stress measured by Parental Stress Index-Short Form (PSI-SF: score ranges from 15% to 100% with higher scores indicating more stress) at baseline, after 5 days, after 9 days and after 28 days of intervention.
Parental quality of life | 0-4 weeks
  Difference in parental quality of life measured by World Health Organization Quality Of Life questionnaire - short version (WHOQOL-BREF: score ranges from 0 to 100 with higher scores indicating better quality of life ) at baseline, after 5 days, after 9 days and after 28 days of intervention.
Weight | 0-4 weeks
  Difference in weight (grams) at baseline, after 14 days and after 28 days of intervention.
Length | 0-4 weeks
  Difference in length (cm) at baseline, after 14 days and after 28 days of intervention.
Weight-for-age | 0-4 weeks
  Difference in weight-for-age z-scores calculated using the World Health Organization Child Growth Standards at baseline, after 14 days and after 28 days of intervention.
Length-for-age | 0-4 weeks
  Difference in length-for-age z-scores calculated using the World Health Organization Child Growth Standards at baseline, after 14 days and after 28 days of intervention.
Weight-for-length | 0-4 weeks
  Difference in weight-for-length z-scores calculated using the World Health Organization Child Growth Standards at baseline, after 14 days and after 28 days of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro López-Escobar, Dr., Principal Investigator — Hospital Universitario General de Villalba
Locations (1):
- HM hospitales, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No